CLINICAL TRIAL: NCT04254432
Title: Safety and Feasibility of Remote Ischemic Conditioning on Prehypertension and Early-Stage Hypertension
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, vice president, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIC-HP-1
Record Dates: First submitted 2020-01-22; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Prehypertension; Remote Ischemic Conditioning; Early Stage Hypertension
Keywords: hypertension; remote ischemic conditioning
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- remote ischemic conditioning arm (Experimental): Device: remote ischemic conditioningRIC is a physical strategy performed by an electric auto-control device with cuffs placed on unilateral arms and inflated to 200 mmHg for 5-min followed by deflation for 5-min, the procedures are performed repeatedly for 5 times# two times per day. The duration of the treatment is 30+/-2days. Other Names:• RICDevice: ambulatory blood pressure monitoring diagnostic technique for measuring blood pressure in daily life by means of automatic intermittent timing. Because ABPM has overcome the limitations of clinic blood pressure measurement, observation error and white coat effect, it can objectively reflect the actual level and fluctuation of blood pressure. Each patient of the two arms will use ABPM measure blood pressure before and after RIC or sham RIC treatment
  Interventions: Device: remote ischemic conditioning

INTERVENTIONS:
Device: remote ischemic conditioning — RIC is a physical strategy performed by an electric auto-control device with cuffs placed on unilateral arms and inflated to 200 mmHg for 5-min followed by deflation for 5-min, the procedures are performed repeatedly for 5 times# two times per day. The duration of the treatment is 4 weeks.

SUMMARY:
Nowadays, the incidence of stroke in China has reached 1.6‰, and this disease has become a primary cause of death in China. One of its major risk factors is hypertension. As shown in the researches, the risk of stroke grows remarkably when the blood pressure increases and there exists a log-linear relationship between them. Systolic pressure and diastolic pressure relate to the risk of stroke independently. Systolic pressure decreasing 10mmHg will reduce the stroke risk by 31% and a decrease of 1~3mmHg will reduce the stroke risk by20~30%. As to diastolic pressure, a 5mmHg decrease will reduce the stroke risk by 34% and a 10mmHg decrease will reduce the stroke risk by 56%.In addition, patients with isolated systolic hypertension (SPB≥160mmHg, DPB≤90mmHg) or critical isolated systolic hypertension (SPB=140~159mmHg, DPB< 90mmHg) will suffer a higher risk of stroke than people with normal blood pressure. The ACC has already revised its Hypertension ManagementGuidelines of the standard of diagnosis for hypertension and the timing of starting medical treatment in hypertensive patients. Because more and more researches shown that people with blood pressure between 120-139/80-89mmHg have higher risk of ASCVSD compared to those with blood pressure lower than120/80mmHg; However, in China, the diagnostic criteria for hypertension has not been revised yet. Therefore, we still have a blind spot in treating such patients who suffer from borderline systolic hypertension at 130~140 mmHg of blood-pressure with or without ASCVD or those with the first stage hypertension but refusing to take anti-hypertension drugs. What is more, most of them are middle-aged adults, once they have a stroke, it would lead to terrible and costly consequences to both their family and society. Thus, it is necessary to explore new non-pharmacological methods to control blood pressure for reducing the risk of stroke

ELIGIBILITY:
Inclusion Criteria:

* systolic blood pressure between 160 and 125 mmHg or diastolic blood pressure between 80 and 100 mmHg
* age≥18
* essential hypertension
* patient did not take anti-hypertensive medicine regularly

Exclusion Criteria:

* patients with severe uncontrolled diabetes
* contraindication for remote ischemic preconditioning
* life expectancy less than 1 year
* patients with atrial fibrillation or other kind of arrhythmia
* unwilling to be followed up or poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
tolerability and feasibility of remote ischemic conditioning on hypertension | 4 weeks
  there are 56 treatments in totall during 4weeks， the percentage of the completement of each treatment would be used to mearure the tolerance.

SECONDARY OUTCOMES:
safety of remote ischemic conditioning on hypertension | 4 weeks
  all the adverse effect would be recorded and the percetage of adverse effect happened in the group would be used to measure the safety.

OTHER OUTCOMES:
clinical efficacy of remote ischemic conditioning on hyperetension | 4 weeks
  the systolic blood pressure and diastolic blood pressure before and after the treatment would be recorded. the defference between baseline BP and that after treatment would be used to measure efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes